CLINICAL TRIAL: NCT00266526
Title: A Bicentre Open Label Randomised Pilot Study for Proof of Safety and Efficacy of Immunotherapy With an Aluminium Hydroxide-adsorbed Recombinant Hypoallergenic Derivative of the Major Birch Pollen Allergen Bet v 1-FV Versus a Depot Extract of Natural Birch Allergen
Brief Title: Specific Immunotherapy With Recombinant Birch Pollen Allergen rBet v1-FV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Al0303rB
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Birch Pollen Allergy
Keywords: Allergy; Birch pollen; Recombinant
MeSH Terms: conditions — Hypersensitivity

INTERVENTIONS:
Biological: Recombinant birch pollen

SUMMARY:
Specific immunotherapy with recombinant birch pollen allergen rBet v1-FV

ELIGIBILITY:
Inclusion Criteria:

* Positive RAST result to birch pollen
* Positive Skin Prick Test reaction to birch pollen
* positive nasal provocation test result to birch pollen extract

Exclusion Criteria:

* serious chronic diseases
* other relevant seasonal allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2003-07; Primary Completion 2004-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Narkus, M.D., Principal Investigator
Locations (1):
- Allergopharma GmbH & Co. KG, Reinbek, Germany

REFERENCES:
- [Derived] Klimek L, Bachert C, Lukat KF, Pfaar O, Meyer H, Narkus A. Allergy immunotherapy with a hypoallergenic recombinant birch pollen allergen rBet v 1-FV in a randomized controlled trial. Clin Transl Allergy. 2015 Aug 3;5:28. doi: 10.1186/s13601-015-0071-x. eCollection 2015. PMID 26328056
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de